CLINICAL TRIAL: NCT06304649
Title: Clinical Evaluation of Cast21 Short Arm Product During Treatment of Distal Radial or Distal Ulnar Fractures
Acronym: Cast21 SAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cast21 (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cast21CHLA2023Study1SAP
Record Dates: First submitted 2023-12-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Fractures, Closed; Fractures Bone; Fracture; Fractures; Radius; Fracture, Lower or Distal End; Ulna Fractures; Radius Distal Fracture
MeSH Terms: conditions — Fractures, Closed; Fractures, Bone; Ulna Fractures; Wrist Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cast21 Short Arm Product (Experimental)
  Interventions: Device: Cast or brace alternative

INTERVENTIONS:
Device: Cast or brace alternative — Waterproof alternative to a cast or brace for broken bones

SUMMARY:
The primary objective of this study will be the collection of preliminary clinical evidence to indicate that Cast21 Short Arm Product is no worse than the current standard of care arm immobilization devices in pediatric patients.

A secondary objective will be to characterize the clinician and patient experience with the Cast21 Short Arm Product.

ELIGIBILITY:
Inclusion Criteria:

* Demographic characteristics: all persons ages 3 and above, regardless of the race and sex will be eligible to participate in this study
* Medical condition: participants must present with a closed, nondisplaced, or minimally displaced distal radius fracture and/or distal ulnar fracture that does not require a bone reduction procedure within 10 days from the date of injury
* Sizing: participants eligible for the Cast21 Short Arm Product must undergo sizing conducted by the clinical staff to ensure fit into one of the products (sizes XS-L)

Exclusion Criteria:

* Participants requiring a surgical intervention
* Participants with moderately displaced or angulated fractures or fractures requiring a bone reduction procedure.
* Participants with a known history of bone diseases e.g. osteogenesis imperfecta or other pathologic bone conditions
* Participants with pathologic fractures e.g., presence of bone cyst
* Participants who smoke
* Participants with pre-existing skin infection or condition of the lower arm (participants exhibiting only minor skin abrasions, lacerations, or skin condition might be eligible per clinical investigator's discretion)

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical determination of healing (standard of care) | At treatment completion, an average of 4 weeks
  A binary determination of healing after the intervention will be asserted by the clinician
Range of Motion (standard of care) | At treatment completion, an average of 4 weeks
  Clinicians will asses patients for a binary determination of Full Range of Motion or Limited Range of Motion

SECONDARY OUTCOMES:
Patient Reported Outcomes - Pain | Before treatment (0 Days) and at treatment completion, an average of 4 weeks
  Patient pain scores with the Wong-Baker FACES Pain Rating Scale will be assessed. The rating scale is 1 (min) to 10 (max) with lower scores being a better outcome.
Patient Reported Outcomes - Satisfaction | At treatment completion, an average of 4 weeks
  A questionnaire adapted from the Patient-Reported Outcomes Measurement Information System (PROMIS) scale will be administered. The scale is 1 (min) to 5 (max), with high scores indicating a better outcome.
Physical Therapy Referral | At treatment completion, an average of 4 weeks
  A binary referral to physical therapy as part of the standard of care will be observed if the patient's range of motion (see Primary Outcome 2) is such that the clinician will refer more care.